CLINICAL TRIAL: NCT02935127
Title: Absorbable Sutures in Peripheral Vascular Surgery
Brief Title: Absorbable Sutures in Vascular Surgery
Acronym: ASPeVaS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Professor, University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ER.ALL.2016.02
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Peripheral Vascular Disease
Keywords: absorbable sutures
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absorbable Group (Experimental): In this group of patients absorbable sutures will be used for vascular anastomoses.
  Interventions: Procedure: Absorbable suture
- Non-Absorbable Group (Experimental): In this group of patients non-absorbable sutures will be used for vascular anastomoses.
  Interventions: Procedure: Non-Absorbable suture

INTERVENTIONS:
Procedure: Absorbable suture — Vascular anastomoses will be performed with absorbable materials
  Arms: Absorbable Group
Procedure: Non-Absorbable suture — Vascular anastomoses will be performed with non-absorbable materials
  Arms: Non-Absorbable Group

SUMMARY:
Absorbable sutures are not generally accepted by the majority of vascular surgeons for the possible complications such as the breakage of the suture at the anastomoses level. Some experimental and clinical studies in the current literature demonstrated that the use of absorbable sutures may even reduce some important complications such as restenosis.

The aim of this study is to compare absorbable and non-absorbable sutures in patients undergoing peripheral vascular surgery with vein bypass grafting.

DETAILED DESCRIPTION:
Infrainguinal vein graft procedures may be performed, generally, on patients with critical limb ischemia (CLI) or popliteal artery aneurysm (PAA). Autologous vein graft, when adequate and available, is usually the preferred conduit, especially in the below knee vascular districts. Vein grafts may complicate with the onset of stenoses (up to 30% of cases). Such complications may develop, due to myointimal hyperplasia along the body of the graft or, more often, at the proximal or distal anastomoses where sutures are performed. In vascular surgery procedures, in case of arterial anastomoses, absorbable suture material is generally not preferred, mainly for the fear of breakage of the suture line. Previous experimental studies performed in animals and humans and a recent clinical study performed in humans on carotid surgery showed that absorbable sutures used in vascular surgery may even reduce the development of intimal hyperplasia and may reduce postoperative stenotic complications. The aim of this study is to evaluate the early and long-term results of absorbable sutures used in peripheral vascular surgery.

This is an open-label, parallel group study.

Patients undergoing vein bass grafting for CLI or PAA may be suitable for entry into ASPeVas trial. They must satisfy the following inclusion criteria:

Both sex. Age > 18 years old. Patients undergoing femoropopliteal or femorodistal vein bypass grafting; must be able to give informed consent; have no significant co-morbidity that makes life expectancy less than six months.

The randomisation process consists as follows: once a patient have consented entering the trial, an envelop is opened and the patient is offered the type of suture (absorbable or non absorbable) regardless of the surgical technique which is going to be performed (femoropopliteal or femorodistal vein bypass grafting).

All patients have to be followed-up, the day after the operation (time 0) and then subsequently at 1, 3,6,9,12 and 18 months.

At each appointment, Ankle Brachial Pressure Index (ABPI) is measured and then Duplex scanning (DS) is performed. In particular, by means of DS the peak systolic flow velocity (PSFV) at multiple sites along the entire graft is measured. A graft at risk of failure was defined as having a PSFV < 45 cm/s or a ratio of V2 (peak velocity at the site of the stenosis) to V1 (peak systolic velocity at any other point within 2 cm at the normal adjacent graft) > 2. Any other irregularities, such as inflow/outflow problems, graft dilatation will be also recorded.

Clinical signs of a failing graft will be collected: disabling claudication, ischemic pain, ischemic ulcers.

ELIGIBILITY:
inclusion criteria:

* Patients undergoing femoropopliteal or femorodistal vein bypass grafting;
* Patients able to give informed consent;
* Patients having no significant co-morbidity that makes life expectancy less than six months.

exclusion criteria:

* patients that do not meet the aforementioned criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Flow Velocity in the graft | 18 months
  centimeters per second (cm/sec)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D., PhD., Principal Investigator — University Magna Graecia of Catanzaro; Stefano de Franciscis, M.D., Study Chair — University Magna Graecia of Catanzaro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gasbarro V, Traina L, Mascoli F, Coscia V, Buffone G, Grande R, Fugetto F, Butrico L, de Franciscis S, Serra R. Absorbable suture material in carotid surgery. Vasa. 2015 Nov;44(6):451-7. doi: 10.1024/0301-1526/a000468. PMID 26515222